CLINICAL TRIAL: NCT04118712
Title: Pediatric Ovarian Tissue Banking - Operative Specimens From Females 0-18 Years of Age
Acronym: OTB
Status: Recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-726
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Benign Cysts Ovarian; Cystectomy; Torsion; Malignant Cysts Ovarian

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — ovarian tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A child is eligible to participate in this study because she is having surgery on her ovary. The investigators may obtain a sample of any discarded tissue from the surgery for an ovarian tissue library. This study is being conducted to understand how common ovarian conditions effect the number and quality of ovarian follicles and the reproductive potential of the ovary.

DETAILED DESCRIPTION:
The investigators intend to enroll 100 girls and women in this study who are undergoing surgery involving the ovary. This may include patients with different conditions for comparison, such as ovarian cysts or masses and ovarian torsion. For each patient, the investigators will obtain the discarded tissue from the operating room after the affected ovarian tissue is resected. The tissue sample will only be taken for the tissue library from ovarian tissue that would otherwise be discarded.

No additional tissue will be collected other than that which is already removed as part of the ovarian procedure. No additional surgery or other procedures will be performed for the purposes of this study. The tissue will be assigned a study ID number and the age, gender and diagnosis of the child will be entered on the tissue library log and maintained for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Pre and Post Pubertal females
* Ages 0-18 years old
* Undergoing scheduled or emergent operative procedures involving the ovary

  1. oophorectomy (torsion, benign mass/cyst, malignant mass/cyst)
  2. ovarian cystectomy

Exclusion Criteria:

* Pregnant females

Max Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Patient recruitment could occur in either the pediatric surgery outpatient clinic or during hospital admission depending on the underlying condition and urgency of the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10-18 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Ovarian Tissue Banking | October 2016- December 2030
  The primary purpose of this study is analyzing the histologically ovarian tissue obtained surgically due to different ovarian pathologies. The tissue will be stained and follicles of varying stages will be counted and compared for different patient ages and ovarian pathologies. The extra-cellular matrix will also be stained and compared between different patient ages and ovarian pathologies.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rowell, MD, Study Director — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Childrens Hospital, Chicago, Illinois, United States